CLINICAL TRIAL: NCT06222385
Title: Measuring and Monitoring Brain Health in Older Adults: The Applied Cognition Glymphatic Function Study at The Villages
Brief Title: Applied Cognition Benchmarking Study
Acronym: BRAIN3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Cognition (Industry)
Collaborators: University of Florida Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: AC.2022.02
Record Dates: First submitted 2024-01-04; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Cross-over randomized study
Who Masked: Outcomes Assessor
Masking Description: Visit type was masked to neuroimaging assessors and blood biomarker analysis laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sleep Opportunity-Sleep Deprivation (Experimental): Participant randomized to overnight sleep period with a morning wake period on first visit of cross-over study.
  Interventions: Diagnostic Test: Device measurements during overnight sleep and morning wake
- Sleep Deprivation-Sleep Opportunity (Experimental): Participant randomized to overnight sleep deprivation period with a morning recovery sleep period on first visit of cross-over study.
  Interventions: Diagnostic Test: Device measurements during overnight wake and morning sleep

INTERVENTIONS:
Diagnostic Test: Device measurements during overnight sleep and morning wake — Overnight period and morning period device measurements
  Arms: Sleep Opportunity-Sleep Deprivation
Diagnostic Test: Device measurements during overnight wake and morning sleep — Overnight period and morning period device measurements
  Arms: Sleep Deprivation-Sleep Opportunity

SUMMARY:
This is a cross-over randomized study to validate the Sponsor investigational medical device against measurements of glymphatic function from MRI-based neuroimaging, EEG, blood biomarkers and cognitive tests in healthy older volunteers.

DETAILED DESCRIPTION:
The study population will consist of healthy individuals, ages 55 to 65, that are cognitively normal and do not have a medical history of neurological or sleep disorder, cardiovascular disease, hypertension, or diabetes. The objectives of this study are to define whether sleep- and wake-associated device measurements (i) faithfully reflect glymphatic function measured by gold-standard contrast enhanced MRI and non-invasive MRI-based measures of glymphatic function; (ii) replicate pre-clinical findings between sleep EEG power bands and glymphatic flow; (iii) predict plasma levels of Alzheimer's disease (AD)-related biomarkers; and (iv) predict morning cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a Montreal Cognitive Assessment (MoCA) score at least 26.
2. Participants must have a Geriatric Depression Scale (GDS) 15-item score of 4 or less.

Exclusion Criteria:

1. Participants with a formal diagnosis of any sleep disorder (e.g., sleep apnea on positive-airway-pressure (PAP) therapy, insomnia, restless leg syndrome, circadian rhythm sleep disorder, parasomnia).
2. Participants with a history of significant neurological disease or history of epilepsy.
3. Participants with cardiovascular disease or cardiovascular risk factors (smoking or hypertension).
4. Participants with diabetes.
5. Participants with traumatic brain injury, or serious mental illness including bipolar disorder, schizophrenia, major depressive disorder or post-traumatic stress disorder.
6. Participants who have taken in the past 30 days prescribed or overthe- counter (OTC) stimulants, sleeping medications, or psychiatric medications including antidepressants.
7. Participants who consume more than 400 mg/day of caffeine. Participants will be required to not consume caffeine beginning 12pm on the day-of the sleep study.
8. Female Participants who consume more than 3 alcoholic drinks on any day or more than 7 drinks per week. Male participants who consume more than 4 alcoholic drinks on any day or more than 14 drinks per week.
9. Participants planning travel to alternate time zones within two weeks of study participation
10. Participants with travel plans or conflicts that would prevent them from either Study Visit.
11. Participants who are enrolled in other research studies and are receiving an investigational drug within 30 days of the planned start date.
12. Participants who have any condition that, in the opinion of the Sponsor Principal Investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements.
13. Participants with absolute or relative contraindications to MRI imaging based on current up-to-date screening questionnaires including claustrophobia, inability to lie still on their back for 30-45 minutes or require sedation prior to the MRI.
14. Participants with a head circumference greater than 60 cm that would prevent use of a high-resolution 64 channel MRI head coil required for this study
15. Participants who have a pre-planned surgery or medical procedure that would interfere with the conduct of the study.
16. Participants who have an implanted medical device or contraindications that would exclude MRIs
17. Participants with a serious infection requiring medical attention in the past 30 days
18. Participants with a diagnosis of substance use-disorder in the past 2 years.
19. Participants with known acute or chronic kidney disease and/or compromised GFR.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Contrast-enhanced MRI | Immediately after the overnight sleep/wake period
  Overnight sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic function measured by ROI parenchymal signal intensity using gold-standard contrast-enhanced MRI for gray and white matter ROI.
Non-invasive MRI - diffusion-based intravoxel incoherent motion | Immediately before and immediately after each sleep/wake period
  Sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic function measured by non-invasive MRI measures of glymphatic function using diffusion-based intravoxel incoherent motion (IVIM)-MRI (long-distance water transport) (diffusion signal, a.u.).
Non-invasive MRI - fast functional MRI | Immediately before and immediately after each sleep/wake period
  Sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic function measured by non-invasive MRI measures of glymphatic function using fast functional MRI (f-MRI) low-frequency vasomotor oscillations, Hz.
Non-invasive MRI - T1/FLAIR-based assessment | Immediately before and immediately after each sleep/wake period
  Sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic function measured by non-invasive MRI measures of glymphatic function using T1/FLAIR-based assessment of MRI-visible perivascular spaces (MVPVS) that are structural indicators of perivascular impairment, (a.u.).
Non-invasive MRI - multi-echo arterial spin-labeling | Immediately before and immediately after each sleep/wake period
  Sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic function measured by non-invasive MRI measures of glymphatic function using multi-echo arterial spin-labeling (ME-ASL)-MRI (glial-vascular water transport) (flow in ml/sec).
Non-invasive MRI - phase-contrast | Immediately before and immediately after each sleep/wake period
  Sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic function measured by non-invasive MRI measures of glymphatic function using phase-contrast (PC)-MRI (aqueductal cerebral spinal fluid (CSF) flow) (flow in ml/sec).

SECONDARY OUTCOMES:
Sleep EEG | Measurements sampled every 5 to 10 minutes during the overnight sleep period
  Device overnight sleep measurements (impedances in milli-ohms) correlations with overnight recorded sleep EEG power bands (relative delta, theta, alpha and beta power in %) and heart rate replicate pre-clinical correlations of glymphatic flow (measured using 2-photon microscopy in a.u.) with EEG power bands (relative delta, theta, alpha and beta power in %) and heart rate.
Blood biomarkers | Immediately before and immediately after each sleep/wake period
  Sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic clearance measured by amyloid beta40, beta42, n-tau 181, n-tau 217, p-tau 181, p-tau 217 blood biomarkers
Cognitive function - trail making tests A&B | Immediately after the sleep/wake period
  Overnight sleep- and wake-associated device measurements predict morning cognitive performance based on Trail Making Tests A&B (time in seconds).
Cognitive function - symbol digit modality test | Immediately after the sleep/wake period
  Overnight sleep- and wake-associated device measurements predict morning cognitive performance based on symbol digit modality test (SDMT) (number correct).
Cognitive function - psychomotor vigilance test | Immediately after the sleep/wake period
  Overnight sleep- and wake-associated device measurements predict morning cognitive performance based on psychomotor vigilance test (PVT) (mean and standard deviation of reaction time).
Cognitive function - digits forward recall | Immediately after the sleep/wake period
  Overnight sleep- and wake-associated device measurements predict morning cognitive performance based on digits forward recall (maximum number of correctly recalled digits).

CONTACTS AND LOCATIONS:
Overall Officials: Carla Vandeweerd, PhD, Principal Investigator — UF Health
Locations (1):
- UF Health - Precision Health Research Center, The Villages, Florida, United States